CLINICAL TRIAL: NCT06167759
Title: Preventing Opioid Misuse Through Safe Opioid Use Agreements Between Patients and Surgical Providers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Jonah Stulberg, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HSC-MS-22-0807
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Opioid Use; Inguinal Hernia; Ventral Hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Use Agreement (Experimental): Patients in this group will be administered a safe opioid use agreement by the research coordinator. This agreement is in addition to any routine education and counseling provided by the surgical team.
  Interventions: Other: Opioid Use Agreement
- Standard of Care (No Intervention): Patients in this group will receive standard care which includes safe opioid education from the surgical care team.

INTERVENTIONS:
Other: Opioid Use Agreement — This was previously developed specifically for surgical patients using a modified Delphi method with a group of experts (including surgeons, nurses, advanced practices providers, quality improvement experts, and patients).
  Arms: Opioid Use Agreement

SUMMARY:
The effect of pain agreements to reduce opioid misuse is an accepted practice in many settings, but it has never been applied to the acute care setting. Pain agreements are considered the standard of care for chronic pain management reliant on opioid prescribing, and they are a mandated component of care in many states. Therefore, the adjunct of safe opioid use agreements into acute pain management offers a logical extension of current practices from chronic pain management.

This study will test the use of agreements to improve safe opioid use to prevent misuse and opioid-related harm.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (at least 18 years of age), of any gender, who speak English or Spanish, undergoing general surgery procedures with a high likelihood of receiving an opioid prescription (bariatric, inguinal hernia, or ventral hernia), who have their preoperative appointment at UT Physicians Health Center at Memorial Hermann Sugar Land Medical Plaza, Lyndon Baines Johnson, and Bellaire

Exclusion Criteria:

Patients with a known allergy or contra-indication to opioids, pregnancy, signification cognitive impairment, history of opioid misuse/abuse, chronic opioid use, readmission before the follow up appointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient self-reported disposal of prescription opioids | 25-40 days after surgery
  Patient self-reported disposal of prescription opioids

SECONDARY OUTCOMES:
Opioid pills used | 25-40 days after surgery
  Number of opioid pill used if opioid prescription was filled
Opioid pills leftover | 25-40 days after surgery
  Number of opioid pills left over if opioid prescription was filled
Storage method | 25-40 days after surgery
  If opioid prescription was filled, how the opioid pills were stored
Disposal method | 25-40 days after surgery
  If opioid prescription was filled, how the opioid pills were disposed
Other pain management strategies | 25-40 days after surgery
  Other pain management strategies that were used

CONTACTS AND LOCATIONS:
Overall Officials: Jonah J Stulberg, MD, Principal Investigator — UTHealth
Locations (3):
- United States (3):
  - UT Physicians-MIST Bellaire Clinic, Bellaire, Texas
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - UT Physicians-MIST Sugar Land Clinic, Sugar Land, Texas